CLINICAL TRIAL: NCT06839885
Title: Evaluation of the Effects of Hydrotherapy on Lower Extremity Volume, Quality of Life, and Functionality in Patients Diagnosed With Unilateral Lower Extremity Lymphedema
Brief Title: Effects of Hydrotherapy on Unilateral Lower Extremity Lymphedema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Çiğdem Aşlı, Medical Doctor, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GaziosmanpasaTREH-FTR-ÇA-001
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Lower Limb Lymphedema; Unilateral Leg Edema
Keywords: Aerobic exercise; Hydrotherapy; Functionality; Gynecological cancer; Lymphedema; Exercise capacity; Quality of life
MeSH Terms: conditions — Lymphedema | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: two groups: an intervention group and a control group
Masking Description: The control group will receive a home exercise program, while the intervention group will receive both a home exercise program and hydrotherapy. Outcome assessments will be conducted by an investigator who is blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Patients with primary or secondary unilateral lower extremity lymphedema who have received at least 2 weeks of Complex Decongestive Therapy in the past year and completed their treatment at least 3 months ago, and who agreed to participate in the study, were included in the study at Health Sciences University Gaziosmanpasa Training and Research Hospital, Department of Physical Medicine and Rehabilitation. Prior to treatment, all patients were planned to receive education about the treatment to be applied in the form of a home program. Patients were planned to be treated in the hydrotherapy unit during lunch breaks under the supervision of a volunteer physiotherapist.
  After the initial assessments, patients in the control group will receive a home exercise program and self-drainage.
  Interventions: Other: Control group
- Intervention Group (Experimental): Patients with primary or secondary unilateral lower extremity lymphedema who have received at least 2 weeks of Complex Decongestive Therapy in the last year and completed treatment at least 3 months ago, and who agreed to participate in the study, were included in the study at Health Sciences University Gaziosmanpasa Training and Research Hospital, Department of Physical Medicine and Rehabilitation. Prior to treatment, all patients were planned to receive education about the treatment to be applied in the form of a home program. The patients were planned to be treated in the hydrotherapy unit during lunch breaks, under the supervision of a volunteer physiotherapist.
  After the initial assessments, patients in the study group will perform aquatic exercises in groups of 5 or 7 participants, three times a week for 6 weeks, under the supervision of a physiotherapist. Patients in the intervention group will receive a home exercise program and self-drainage.
  Interventions: Other: Interventional group

INTERVENTIONS:
Other: Interventional group — Patients with primary or secondary unilateral lower extremity lymphedema who have received at least 2 weeks of Complex Decongestive Therapy in the last year and completed treatment at least 3 months ago, and who agreed to participate in the study, were included in the study at Health Sciences University Gaziosmanpasa Training and Research Hospital, Department of Physical Medicine and Rehabilitation. Prior to treatment, all patients were planned to receive education about the treatment to be applied in the form of a home program. The patients were planned to be treated in the hydrotherapy unit during lunch breaks, under the supervision of a volunteer physiotherapist.
  After the initial assessments, patients in the study group will perform aquatic exercises in groups of 5 or 7 participants, three times a week for 6 weeks, under the supervision of a physiotherapist.Patients in the intervention group will receive a home exercise program and self-drainage.
  Arms: Intervention Group
Other: Control group — Patients with primary or secondary unilateral lower extremity lymphedema who have received at least 2 weeks of Complex Decongestive Therapy in the past year and completed their treatment at least 3 months ago, and who agreed to participate in the study, were included in the study at Health Sciences University Gaziosmanpasa Training and Research Hospital, Department of Physical Medicine and Rehabilitation. Prior to treatment, all patients were planned to receive education about the treatment to be applied in the form of a home program. Patients were planned to be treated in the hydrotherapy unit during lunch breaks under the supervision of a volunteer physiotherapist.
  After the initial assessments, patients in the control group will receive a home exercise program and self-drainage.
  Arms: Control group

SUMMARY:
Lymphedema is a chronic condition that negatively affects patients' quality of life and lower extremity functions, causing swelling and a feeling of heaviness in the extremity, as well as posing an economic burden. The gold standard in lymphedema treatment is complex decongestive therapy.Manual lymphatic drainage, skin care, the use of compression garments, and home exercise programs play an important role. Exercise therapies lead to a reduction in volume and an improvement in functionality and quality of life in patients with lymphedema. However, studies on this subject have mostly focused on upper extremity lymphedema. This study aims to compare the effects of a home exercise program and hydrotherapy combined with a home exercise program on quality of life, lower extremity functionality, exercise capacity, and edema severity in patients with unilateral lower extremity lymphedema

DETAILED DESCRIPTION:
This study included patients, with in the control group and in the intervention group, who applied to the lymphedema outpatient clinic at Health Sciences University Gaziosmanpasa Training and Research Hospital, Department of Physical Therapy and Rehabilitation. The demographic and clinical data of the patients were recorded. Before treatment, limb volume was assessed using the circumference measurement method, quality of life was evaluated with the Lymphedema Quality of Life Questionnaire (LYMQOL), lower extremity functionality was assessed with the Lower Extremity Functional Scale (LEFS), and exercise capacity was measured using the 10-Meter Walk Test. Patients in the control group followed only a home exercise program for 6 weeks, while the intervention group received hydrotherapy combined with a home exercise program for the same period. Hydrotherapy was conducted as 30-minute aquatic exercise sessions in groups of 5-7 participants, in a hydrotherapy pool with a depth of 130 cm and a temperature of 30-31°C, under the supervision of a trained physiotherapist. At the end of the treatment, patients were re-evaluated in terms of volume, functionality, quality of life, and exercise capacity. The two groups were compared regarding volume measurement, functionality, and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary or secondary unilateral lower extremity lymphedema diagnosis
* Patients who have received at least 2 weeks of complex decongestive therapy in the past
* Patients who are cooperative with hydrotherapy treatments
* Patients who are willing to participate in the treatment
* Patients aged 18-75

Exclusion Criteria:

* Patients who are unable to perform the evaluation parameters
* Patients with serious systemic diseases that may prevent exercise
* Patients who have had an injury and/or surgery in the last 6 months
* Conditions where hydrotherapy is contraindicated (severe fear of water, behavioral problems, shortness of breath at rest, incontinence, known chlorine allergy, open wound, acute systemic illness, epilepsy, tracheostomy, permanent drain, immunodeficiency)
* Patients with an active infection anywhere in the body
* Patients who have undergone sentinel lymph node biopsy
* Patients with active metastatic disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Volume measurement | six weeks
  Patients who applied to the lymphedema outpatient clinic had their leg circumference measurements taken before starting the treatment program and 6 weeks later, starting from the ankle (medial malleolus) and at 4 cm intervals up to the inguinal region. Using these measured data, an approximate volume calculation was made using the circumference (Frustum) method.

SECONDARY OUTCOMES:
Lymphedema Quality of Life Questionnaire-Leg( LYMQOL-Leg) | six weeks
  The LYMQOL-leg questionnaire was used to assess the quality of life specific to lymphedema before and after treatment for all patients participating in the study. The questionnaires were administered through face-to-face interviews.
  LYMQOL can be used in clinical assessments for patients with lymphedema, as well as in evaluating treatment outcomes. LYMQOL is a disease-specific quality of life scale for lymphedema patients. The LYMQOL questionnaire has two separate sections for evaluating the upper and lower extremities: LYMQOL-arm and LYMQOL-leg. The questions in the LYMQOL-leg questionnaire are related to 4 sections. This questionnaire consists of a total of 22 questions. Questions 1-3 assess function, questions 4-10 assess body image, questions 11-15 assess symptoms, questions 16-21 assess mood, and question 22 evaluates 'general quality of life.' The first 21 questions are scored on a scale of 1-4 (1 = none, 2 = a little, 3 = quite a bit, 4 = very much).
Lower Extremity Functional Scale | six weeks
  The LEFS scale was used to assess the functional status of the lower extremities before and after treatment for all patients participating in the study. The questionnaires were administered through face-to-face interviews. The LEFS questionnaire, used to assess functional status in patients and consists of a total of 20 questions. Each question in the LEFS questionnaire is scored on a scale of 0 to 4 (0 - Extremely difficult or unable to do, 1 - Quite difficult, 2 - Moderately difficult, 3 - Slightly difficult, 4 - No difficulty). The total score ranges from 0 to 80. In the LEFS questionnaire, an increase in the score indicates an improvement in the patient's functional status. The Turkish reliability and validity of this questionnaire have been demonstrated in studies.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Yılmaz Yalçınkaya, Study Director — Gaziosmanpasa Research and Education Hospital
Locations (1):
- GaziosmanpasaTREH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ali KM, El Gammal ER, Eladl HM. Effect of Aqua Therapy Exercises on Postmastectomy Lymphedema: A Prospective Randomized Controlled Trial. Ann Rehabil Med. 2021 Apr;45(2):131-140. doi: 10.5535/arm.20127. Epub 2021 Apr 14. PMID 33849087
- [Background] Dionne A, Goulet S, Leone M, Comtois AS. Aquatic Exercise Training Outcomes on Functional Capacity, Quality of Life, and Lower Limb Lymphedema: Pilot Study. J Altern Complement Med. 2018 Sep/Oct;24(9-10):1007-1009. doi: 10.1089/acm.2018.0041. PMID 30247973
- [Background] Yeung W, Semciw AI. Aquatic Therapy for People with Lymphedema: A Systematic Review and Meta-analysis. Lymphat Res Biol. 2018 Feb;16(1):9-19. doi: 10.1089/lrb.2016.0056. Epub 2017 Mar 27. PMID 28346851